CLINICAL TRIAL: NCT01887457
Title: PIVOTAL: Pharmacological Individualisation of VOriconazole Therapy for AntifungaL Treatment
Brief Title: Individualisation of Voriconazole Antifungal Therapy Antifungal Therapy
Acronym: PIVOTAL
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Transfer of management of study
Sponsor: Brynn Chappell (Other)
Collaborators: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor-Investigator, Brynn Chappell, Clinical Trials Project Manager, The Christie NHS Foundation Trust
Organization: The Christie NHS Foundation Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13_DOG06_172; 2013-002578-34 (EudraCT Number)
Record Dates: First submitted 2013-06-07; First posted 2013-06-26 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Immunocompromised Patient; Aspergillosis; Fusarium
Keywords: voriconazole; VFEND; individualised; personalised
MeSH Terms: conditions — Aspergillosis | interventions — Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Voriconazole (Experimental): Standard adult Voriconazole (VFEND) Loading (1 hr infusion): 6mg/kg at 1 hour and 12 hours on day 1. Followed by standard maintenance dose 4mg/kg at 1 hour and 12 hours on day 2 (1 hour infusion). Day 3 follows the same schedule, expect the dose is adjusted, this dose is used on Day 4 and a further dose adjustment is made that is administered as above on Day 5.
  Interventions: Drug: VFEND

INTERVENTIONS:
Drug: VFEND — voriconazole will be administered in iv form
  Other Names: voriconazole

SUMMARY:
This is a trial to determine whether giving a patient a tailored dose of voriconazole is safe and effective.

DETAILED DESCRIPTION:
Invasive fungal infections are a major cause of morbidity and mortality in patients with haematological malignancy and haematopoietic stem cell transplantation.

Voriconazole is routinely used as a first-line agent for the treatment of invasive aspergillosis, invasive fusariosis and scedosporiosis. Voriconazole has extreme pharmacokinetic variability. Adult patients with a trough concentration of < 1 mg/L have a lower probability of clinical response whereas patients with trough concentrations > 6 mg/L a higher probability of toxicity.

Therapeutic drug monitoring for dose adjustment is advocated but there are no algorithms that enable voriconazole dosage to be reliably adjusted to achieve desired trough concentrations in a timely and optimally precise manner.

Novel ways to deliver optimised antifungal therapy are urgently required and this trial will evaluate whether giving a patients a tailored dose of voriconazole is safe and effective.

Plasma concentrations will be taken in real time and inputted in dose software that will calculate an optimum dose for the required trough concentration of 1-3 mg/L.

The software has been developed using data from phase I and III trials of voriconazole.

ELIGIBILITY:
Inclusion Criteria:

* Any adult ≥18 years old
* Patients where a new course of voriconazole is indicated for suspected or confirmed invasive aspergillosis or other serious fungal infections that is deemed by the treating physician to be susceptible to voriconazole
* Patients must have venous access to permit the administration of voriconazole and enable the procurement of multiple plasma samples to measure voriconazole concentrations.
* Estimated creatinine clearance ≥ 50 mL/min
* Able to give written informed consent
* Considered fit to receive the trial treatment
* Able to remain in the hospital for at least 5 days or until they complete their trial treatment
* Female patients must satisfy the investigator that they are not pregnant, or are not of childbearing potential, or are using adequate contraception
* Men must also use adequate contraception

Exclusion Criteria:

* Patients with an estimated creatinine clearance < 50 mL/minute (this precludes the use of intravenous voriconazole)
* Patients receiving any form of renal replacement therapy i.e. haemodialysis or haemofiltration
* Patients with hepatic insufficiency
* Female patients that are pregnant, breast feeding or planning pregnancy during the study
* Past history of intolerance to voriconazole
* Age <18
* Evidence of a clinically relevant fungal isolate that is resistant to voriconazole
* QT prolongation on ECG
* Use of other medications that contraindicate the use of voriconazole
* Patients receiving any other medications that are contraindicated with the use of voriconazole i.e. terfenadine, long acting barbiturates, ergot alkaloids, etc. (Refer to SMPC). Only patients on rifampicin, rifabutin, phenytoin, and carbamazepine would have voriconazole precluded. Voriconazole influences with the pharmacokinetics of many additional agents- (see SMPC)- most importantly anti-rejection compounds- cyclosporine, tacrolimus]
* Uncontrolled cardiac, respiratory or other disease or any serious medical or psychiatric disorder that would preclude trial therapy or informed consent.
* Hypersensitivity to Voriconazole, its excipients or other triazoles

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Dose adjustment success | Day 5 of treatment
  Dose adjustment success will be evaluated by plasma trough concentration on day 5, successful dose adjustment is defined as a trough concentration of 1-3 mg/L of voriconazole.

SECONDARY OUTCOMES:
Mortality of patients | 35 Day after starting treatment
  To examine the mortality of patients receiving individualised voriconazole dosing
Toxicity | Day 5 of treatment and 35 day follow-up
  To evaluate the adverse events that are attributable to voriconazole as assessed by CTCAE v4.

CONTACTS AND LOCATIONS:
Overall Officials: William Hope, Study Chair — University of Liverpool
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom

REFERENCES:
- See also: Christie NHS website — http://www.christie.nhs.uk/